CLINICAL TRIAL: NCT01569217
Title: Construction of a Database to Identify Early Indicators of Respiratory Muscle Dysfunction in Neuromuscular Patients From the Optoelectronic Plethysmography Assessment of the Thoracoabdominal Motion
Brief Title: Regional Distribution of Ventilation to Assess Respiratory Muscle Dysfunction
Acronym: DREM
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Principal Investigator, Lofaso, MD PhD, Professor, Centre d'Investigation Clinique et Technologique 805
Other Study IDs: 11 003-CCP Ile de France XI; 11.155 bis (Registry Identifier: CCTIRS)
Record Dates: First submitted 2012-03-27; First posted 2012-04-03 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Respiratory Failure; Neuromuscular Disorder; Diaphragmatic Paralysis
Keywords: Diaphragm; Abdomen; Breathing pattern; dyspnea
MeSH Terms: conditions — Respiratory Insufficiency; Neuromuscular Diseases; Respiratory Paralysis; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- respiratory muscle dysfunction patients: Neuromuscular patients
- diaphragmatic dysfunction: patients who present orthopnea, recruitment of accessory muscles, abdominal paradox, respiratory dysfunction or dyssynchronous movement

SUMMARY:
The aim of this study is to better discriminate respiratory muscle dysfunction by comparing the measurements of thoracoabdominal motion obtained by an optoelectronic recording and the conventional tests of respiratory muscle strength. The final objective is to better select in the future the patients who need more specific assessment of diaphragmatic function like "maximal transdiaphragmatic pressure" measurement and "phrenic nerve stimulation".

DETAILED DESCRIPTION:
All patients which had suspected respiratory muscle dysfunction will have usual exploration of the respiratory muscles according to the clinician prescription. These explorations can include :

* Lung volumes in seating and supine position
* Maximal inspiratory and expiratory pressures
* Maximal sniff pressures

And when diaphragmatic dysfunction is suspected :

* Maximal transdiaphragmatic pressure
* Phrenic nerve conduction

These patients will also beneficiate to the determination of volume variations of the upper rib cage, the lower rib cage and the abdominal compartments by using Opto-electronic plethysmography.

ELIGIBILITY:
Inclusion Criteria:

* suspicion of respiratory muscle dysfunction
* indication of diaphragm exploration

Exclusion Criteria:

* acute respiratory failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neuromuscular patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
compartmental distribution of the inspired/expired volumes | 1 hour
  Measurements of the thoraco-abdominal motion and of the global lung volume changes.
  Measurements will be done during spontaneous breathing and during vital capacity maneuvers. Therefore the tidal volume, the inspiratory capacity and the expiratory reserve volume will be measured in liters and for each compartiment (upper thorax, lower thorax, abdomen) contribution of these volumes will be expressed in percentage.

SECONDARY OUTCOMES:
left side and right side contribution to the inspired/expired volumes | 1 hour
  Measurements will be done during spontaneous breathing and during vital capacity maneuvers. Therefore the tidal volume, the inspiratory capacity and the expiratory reserve volume will be measured in liters and each side contribution of these volumes will be expressed in percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Lofaso, MD, PhD, Principal Investigator — Centre d'Investigation Clinique et Technologique 805
Locations (1):
- Raymond Poincaré Hospital, Garches, France